CLINICAL TRIAL: NCT03291418
Title: A Double-Blind, Controlled Study to Compare the Gastrointestinal Safety of a 14-Day Oral Dosing Regimen of ATB-346 to Sodium Naproxen in Healthy Subjects
Brief Title: To Compare the Gastrointestinal Safety of a 14-Day Oral Dosing Regimen of ATB-346 to Sodium Naproxen in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Antibe Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ATB-346-P2GIS
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-09

CONDITIONS: Gastric Ulcer
Keywords: Healthy Volunteers, ATB-346, Naproxen sodium, GI safety
MeSH Terms: conditions — Stomach Ulcer | interventions — 2-(6-methoxy-napthalen-2-yl)-propionic acid 4-thiocarbamoyl-phenyl ester; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Encapsulated tablets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ATB-346 OR Placebo (Experimental): Intervention: Drug: ATB-346 dosed orally at 250 mg once daily for 14 days Intervention: Drug: Placebo (for ATB-346) dosed once daily for 14 days
  Interventions: Drug: ATB-346 OR Placebo
- Naproxen sodium (Active Comparator): Intervention: Drug: naproxen sodium dosed orally at 550 mg twice daily for 14 days
  Interventions: Drug: Naproxen sodium

INTERVENTIONS:
Drug: ATB-346 OR Placebo — Comparison of gastrointestinal effects
  Arms: ATB-346 OR Placebo
Drug: Naproxen sodium — Comparison of gastrointestinal effects
  Other Names: Naprosyn
  Arms: Naproxen sodium

SUMMARY:
A Double-Blind, Controlled Study to Compare the Gastrointestinal Safety of a 14-Day Oral Dosing Regimen of ATB-346 to Sodium Naproxen in Healthy Subjects

DETAILED DESCRIPTION:
Healthy male and female subjects (n=240) are randomized into two dose groups of 120 subjects each. Gastroduodenal endoscopies are performed pre-dose and post-dose, i.e., after 14 days of either ATB-346 (250 mg once daily) or naproxen sodium (550 mg twice daily) and the incidence of gastric mucosal damage is recorded for comparison between the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult subjects ≥18 to ≤65 years of age 2. Healthy subject with no history of significant gastrointestinal (GI) disease, arthritis or bleeding disorders 3. Subject with laboratory values within normal and acceptable ranges or out of range laboratory values deemed non-clinically significant, as per investigator discretion 4. BMI ≤35 kg/m2 5. Non-smoker for >1 month prior to screening 6. Subject able and willing to give written informed consent, and understand and adhere to protocol requirements 7. Female of childbearing potential using adequate birth control for at least 28 days prior to the first dose of the study drug and for 60 days after the last drug administration, as specified in one of the options below:

  * Abstinence from heterosexual intercourse
  * Contraception to include birth control pills, injectable/implant/transdermal patch
  * Intrauterine device
  * Cervical cap or diaphragm with use of spermicide
  * Condom with spermicide Male subjects with female partners of childbearing potential must agree to abstain from sexual intercourse or use on the above forms of contraception for a period of 3 months following the last drug administration.

    8. Female of non-childbearing potential who is either sterile (via complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state for at least one year 9. Subject who consumes no more than 1 alcoholic serving/drink per day (e.g. 355 mL (12 fluid (fl) ounces (oz)) of regular beer; 148 mL (5 fl oz) of wine; 45 mL (1.5 fl oz) of distilled spirits) 10. Subject willing to refrain from alcohol consumption for 48 hours prior to the screening endoscopy and randomization, and 48 hours prior to the Day 14 endoscopy.

    11. Screening endoscopy is free from any observable gastroduodenal erosions or ulcers, and no greater than 10 mucosal petechiae.

Exclusion Criteria:

* 1. Subject with abnormal baseline laboratory values deemed to be clinically significant by the Investigator 2. Ongoing use of any prescription or over-the-counter medications, or natural/herbal or vitamin preparations, that in the opinion of the Investigator would interfere with the study objectives, or impact subject safety (with the exception of systemic contraceptives and hormone replacement therapy) 3. Use of investigational drugs up to thirty (30) days before screening 4. Use of the following medications within two weeks prior to randomization:

  1. NSAIDs, Aspirin, aspirin-containing products or naproxen-containing medications, NSAID-containing products
  2. Proton pump inhibitors
  3. H-2 blockers
  4. Anti-platelet agents
  5. Anti-coagulants
  6. Antimicrobials
  7. Other gastroprotective agents such as antacids, misoprostol, or bismuth-containing products 5. Subject-reported past history of gastrointestinal ulcer or gastrointestinal bleeding, or any clinically significant gastrointestinal disease.

     6. Positive for Helicobacter pylori urea breath test at the screening visit 7. Clinically significant gastrointestinal, hepatic or renal disease, or any other conditions known to significantly impact or interfere with absorption, distribution, metabolism or elimination of the investigational drug(s) 8. Clinically significant past or present diseases or illnesses that, in the opinion of the investigator, would interfere with the study objectives or integrity or with the subject's safety.

     9. Subject with seated pulse rates <50 beats per minute (bpm) or >100 bpm at screening 10. Seated blood pressure <100/60 mm Hg or >140/90 mm Hg at screening 11. Known hypersensitivities to naproxen, other non-steroidal anti-inflammatory (NSAID) agents, related products (including excipients and formulations) 12. Known hypersensitivities to drugs used for sedation during endoscopy 13. Severe hypersensitivity (including angioedema) to any drugs 14. Use of medications with known drug-drug interactions including potent enzyme-modifying drugs, potent inhibitors and/or inducers of CYP enzymes (such as fluoxetine, barbiturates or St. John's Wort) in the previous thirty (30) days before randomization 15. Female who is pregnant or breastfeeding 16. Positive test for HIV antigen/antibody combination, hepatitis B surface antigen (HBsAg), or anti-Hepatitis C virus tests 17. Positive urine drug test at screening 18. Positive urine alcohol test prior to the screening endoscopy 19. Any clinically significant illness up to thirty (30) days before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Gastroduodenal ulcers >=3mm diameter | At completion of 14 days of oral dosing
  Incidence of gastric or duodenal ulcers of at least 3 mm diameter with unequivocal depth

SECONDARY OUTCOMES:
Gastroduodenal ulcers >=5mm diameter | At completion of 14 days of oral dosing
  Incidence of gastric or duodenal ulcers of at least 5 mm diameter with unequivocal depth
gastroduodenal erosions | At completion of 14 days of oral dosing
  Number of gastric and/or duodenal erosions and/or ulcers
Dyspepsia | At completion of 14 days of oral dosing
  Incidence of dyspepsia leading to study withdrawal
Hematocrit | At completion of 14 days of oral dosing
  Change from baseline in hematocrit levels
Thromboxane B2 levels | At completion of 14 days of oral dosing
  Changes from baseline in ex vivo whole blood thromboxane B2 (TXB2) synthesis

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Principal Investigator — Topstone Clinical Research
Locations (1):
- Topstone Clinical Research, Toronto, Ontario, Canada